CLINICAL TRIAL: NCT04221295
Title: PREPARE Trial: a Parallel Arm Multicenter Randomized Trial of Frailty-focused PReoperative Exercise to Decrease PostoperAtive Complications Rates and Disability scorEs
Brief Title: The PREPARE Trial: Exercise Before Surgery to Improve Recovery in Older People With Frailty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190409-01T
Record Dates: First submitted 2019-12-02; First posted 2020-01-09 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Frailty; Surgery--Complications; Disability Physical
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Group allocation will not be indicated in data analyzed by the outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The intervention is a home-based, multimodal exercise prehabilitation program. Exercise is prescribed in one-hour sessions, performed a minimum of three times per week for three weeks, consisting of: 1) strength training, 2) aerobic exercise and 3) flexibility. The intervention group will receive weekly phone calls to gauge adherence, suggest modifications, provide support and track any adverse events.
  Interventions: Behavioral: Exercise Group
- Control Group (No Intervention): The control group will receive the World Health Organization recommendations for physical activity for people greater or equal to the age of 65 years old pamphlet, as well as a guide to healthy eating for older adults.

INTERVENTIONS:
Behavioral: Exercise Group — Previously described in the arm/group descriptions.
  Arms: Exercise Group

SUMMARY:
This study evaluates whether participating in a home-based exercise program leads to lower levels of complication rates and patient-reported disability after surgery. Half of the participants will be randomized into the exercise group, while the other half will be randomized into the control group.

DETAILED DESCRIPTION:
Background: Four out of ten older people having surgery live with frailty, leaving them vulnerable to adverse outcomes due to accumulation of age- and disease-related deficits. An increasing number of people with frailty require surgery. Frailty is associated with a >2-fold increase in complications and new patient-reported disability; absolute rates are >50% and 20% respectively; physical and physiologic deficits are particularly implicated. Mortality, costs and institutionalization after surgery are also significantly associated with frailty.

Despite frailty's strong association with adverse outcomes, few perioperative trials include older people with frailty. Exercise therapy may improve function and decrease complications for other people with frailty by addressing physical and physiologic deficits. However, existing trials are small (median n=54) and single center. Most interventions have been resource-intensive, requiring attendance at hospital-based sessions, which may limit access to many who could benefit. Patient-reported outcomes are also lacking. Therefore, a multicenter trial of home-based exercise therapy before surgery for older people with frailty, powered to address patient-reported outcomes, is needed. Our trial will address these knowledge gaps by testing the effectiveness of home-based preoperative exercise (exercise prehabilitation) in decreasing patient-reported disability and postoperative complications in older people with frailty having major surgery.

Research aims: Estimate the effectiveness of exercise prehabilitation on:

* Co-primary outcomes: patient-reported disability 30-days after surgery and in-hospital complications
* Secondary outcomes: patient-centered (discharge home, survival, 30, 90 and one-year disability scores, quality of life, function) and system-relevant (length of stay, admissions)
* Health economic outcomes: costs, cost-effectiveness

Methods:

Design, setting and participants: Parallel-arm multicenter randomized controlled trial at 11 Canadian hospitals. People => 60 years old with frailty (Clinical Frailty Scale score of 4/9) having major elective non-cardiac surgery (vascular, intrathoracic, intraabdominal, pelvic, ENT) with expected length of stay of => 2 days will be included.

Intervention: Home-based exercise program with demonstrated efficacy, feasibility and acceptability tailored for people with frailty.

Outcomes and sample size: Co-primary outcomes are patient-reported disability 30 days after surgery (validated WHODAS tool) and prospectively collected in-hospital complications (validated POMS tool). 750 participants (375/arm) will provide 98% power for disability (control mean score 35 (SD 25; MID=8)) and 90% power for complications (55% complication rate (25% relative risk reduction)) (α=0.025; 2 pair-wise comparisons).

Due to surgical delays and cancellations as a result of the COVID-19 pandemic, our trial sample size has seen more participants having surgery outside of their expected time to operation than originally predicted. To account for this, and to ensure adequate power for our analyses, our final sample size will be increased to 850 participants.

Expertise: Our team features multidisciplinary clinical and methodological experts, nationally representative knowledge users and patient representatives.

Expected outcomes: Older people with frailty are a growing and vulnerable segment of the surgical population and are under-represented in existing studies. Exercise prehabilitation is a high-priority research question which may be most relevant to people with frailty given their physical and physiologic vulnerabilities. This study, featuring patient-reported outcomes and an integrated knowledge translation approach will produce generalizable findings directly relevant to patients, families, caregivers, and knowledge users.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Elective surgery with expected post-surgery stay of 2 days or more.
* Frailty present (Clinical Frailty Scale (CFS) score of 4/9 or greater)
* Surgery date between 3 and 12 weeks from enrollment

Exclusion Criteria:

* Inability to speak English or French
* Co-morbidity preventing assessment or understanding of questionnaires
* Unable to be contacted by telephone
* Unwilling to participate in exercise program
* Cardiac, neurological or orthopedic procedure
* Palliative surgery
* Certain cardiovascular conditions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital complications | up to 30 days.
  The Postoperative Morbidity Survey (POMS), will be used to define complications. Individuals experiencing any POMS complication or dying in hospital will be said to have experienced a complication.
Patient-reported disability 30 days after surgery | Assessing change in score from baseline data collection to 30 days post-op
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS) will be used . It is a patient-reported disability scale that assesses limitations in six major life domains - cognition, mobility, self-care, social interaction, life activities and participation in society. Participants will report if they have had no difficulty, mild difficulty, moderate difficulty, severe difficulty or extreme difficulty (simply cannot do) with the items listed.

SECONDARY OUTCOMES:
Function - 5 Times Sit to Stand | Assessing change in score from baseline data collection up to 30 days post-op.
  The 5 Times Sit to Stand is a validated test that will be used for measuring the risk of falls and predicting disability in older adults.
Function - Daily and total step count | Assessing the difference in daily and total step count between the exercise group and control group for 30 days post-op.
  Daily and total step counts will be measured, which will predict adverse post-hospitalization outcomes and will reflect physical recovery. They will be recorded daily for the duration of the exercise program (for those in the exercise group) and 30 days after surgery (for all participants) to evaluate functional recovery.
Function - Katz Index of Activities of Daily Living | Assessing change in the participants KATZ ADL score from baseline to post-op day 3, 5, 7 and up to 30 days.
  The Katz Index measures function in activities of daily living (ADL). The ADLs examined are bathing, dressing, toileting, transferring, continence and feeding. If a person is able to perform the ADL independently, they receive 1 point for that activity. If a person is dependent on others to perform the ADL, they receive 0 points for that activity. A score of 6 is high, meaning the person is independent whereas a score of 0 is low, indicating that the person is very dependent.
Function - Falls | Assessing the difference in the occurrence of falls between the exercise group and control group on day 3, 5, 7, up to 30 days, as well as 30-day, 90-day and one-year after surgery.
  Falls will be documented as a way of assessing function.
Health-related quality of life | Assessing any change from baseline to 30, 90 and 365 days post-op.
  EQ-5D EuroQuoL will be used to measure health-related quality of life at baseline, 30, 90 and 365 days after surgery and to inform incremental cost per quality-adjusted life year gained. Participants are asked to select one answer under each domain (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Responses range from having no problems with a particular domain to being unable to engage in that particular domain. Finally, participants are asked to identify on a scale of 0-100 how good or bad their health is on that given day (0 being worst health they can imagine, 100 being best health they can imagine).
All-cause mortality | 30, 90, and 365 days.
  All deaths and death dates will be identified in-hospital or through telephone follow-up.
Health System - Discharge disposition | Up to 30 days post-op.
  Assess where the participant will be discharged to once out of hospital.
Health System - Hospital re-admissions | 30, 90, and 365 days post-op via telephone
  Participants will be asked during the 30 day, 90 day and one-year follow-up calls if they have been readmitted to hospital since hospital discharge.
Health System - Emergency department visits | 365 days post-op
  Emergency department visits since hospital discharge will be captured in the year after surgery
Health System - Long-term care admissions | 30, 90, and 365 days post-op via telephone
  Participants will be asked during the 30 day, 90 day and one-year follow-up calls if they were admitted to a long-term care facility.
Participant Feedback | Participants are asked to reflect on the program during a call the day before surgery.
  A theoretical domains framework participant survey will identify barriers and facilitators to participation in the exercise group. Responses are on a five-point likert scale ranging from "strongly disagree" to "strongly agree", or "never" to "always" depending on the question asked.
Safety (Adverse Events) | Assessing frequency of, or change in any safety events from enrollment up to 30 days post-op in hospital between the exercise group and control group.
  Falls, cardiac or respiratory complications and unplanned healthcare encounters will be collected during the exercise treatment period for the exercise group. For the control group, participants will be asked if they experienced any falls since the time of enrollment up until the day before surgery. Safety data will also be collected should any adverse event take place during any physical assessment data collection time point. Unplanned healthcare encounters will also be collected during the time of enrollment to the day before surgery for the intervention group through chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I McIsaac, MD,MPH,FRCPC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, including data dictionaries, will be available. This includes individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). The Study Protocol, Statistical Analysis Plan and Informed Consent Form will also be made available. Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data. Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to dmcisaac@toh.ca. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to dmcisaac@toh.ca. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.

REFERENCES:
- [Derived] McIsaac DI, Lee S, Fergusson D, Gillis C, Khadaroo RG, Meliambro A, Muscedere J, Eskander A, Moloo H, Nelson G, Saha T, Chun R, Serrano PE, Wijeysundera DN, Taljaard M; PREPARE Trial Investigator Group; Barnes K, Boet S, Boland L, Branje K, Breau R, Bryson GL, Dhalla I, Dixon E, Dobson G, Farnand M, Forster A, Gagne S, Hladkowicz E, Holroyd-Leduc J, Huang A, Hutton J, Jacobsohn E, Joanisse J, Johnson A, Johnson S, Khalil N, Kidd G, Lalu M, Lavallee LT, Le T, Levine M, Love C, McCartney C, McMullen M, Bergamascki LM, Moore R, Mozel M, Nagpal S, Nantel J, Power B, Scheede-Bergdahl C, Tamblyn-Watts L, Thavorn K, Trottier D, van Walraven C, Yang I. Home-Based Prehabilitation for Older Surgical Patients With Frailty: A Randomized Clinical Trial. JAMA Surg. 2025 Dec 3:e255288. doi: 10.1001/jamasurg.2025.5288. Online ahead of print. PMID 41335421
- [Derived] McIsaac DI, Fergusson DA, Khadaroo R, Meliambro A, Muscedere J, Gillis C, Hladkowicz E, Taljaard M; PREPARE Investigators. PREPARE trial: a protocol for a multicentre randomised trial of frailty-focused preoperative exercise to decrease postoperative complication rates and disability scores. BMJ Open. 2022 Aug 8;12(8):e064165. doi: 10.1136/bmjopen-2022-064165. PMID 35940835